CLINICAL TRIAL: NCT06340126
Title: Effects of Active Tissue Release Techniques on Groin Pain, Hip Range of Motion, and Functional Disability in 2nd Trimester of Pregnancy
Brief Title: Effects of Active Tissue Release Techniques on Groin Pain in 2nd Trimester of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0567
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Groin Strain
Keywords: Backache; Pregnancy
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tissue release technique group (Experimental): The group will be treated by active release techniques for 4 weeks, 3 sessions per week. One session will be for 10 minutes. Before each session, an ice pack is applied to the groin area for inflammation if present.
  Interventions: Other: Active release techniques
- Relaxation exercises Group (Active Comparator): Group B will be treated by relaxation exercises only. Relaxation exercises include breathing exercises, pelvic floor exercises, and postural exercises.
  Interventions: Other: Relaxation exercises

INTERVENTIONS:
Other: Active release techniques — Active release techniques are soft tissue systems or movement-based techniques. It is used to treat muscles, nerves, fascia, ligaments, and tendons.
  Arms: active tissue release technique group
Other: Relaxation exercises — Relaxation exercises include breathing exercises, pelvic floor exercises, and postural exercises. Exercises will be done in a sitting position
  Arms: Relaxation exercises Group

SUMMARY:
The study will focus on the effects of active tissue release techniques on groin pain, hip range of motion, and functional disability in 2nd trimester of pregnancy. This will be a randomized controlled trial conducted on 30 participants from Prime Care Hospital. Pregnant women in the second trimester aged between 25 to 35 years, who have groin or round ligament pain will be included in this study. A sample of 30 will be divided into 2 groups. Group A will undergo treatment of active release techniques for 10 minutes thrice a week with no home plan of home relaxation exercises. In contrast, Group B will combine treatment of active release technology with home relaxation exercises. Treatment will be given for 4 weeks and pain will be assessed before and after the treatment through (NPRS) scale. Functional disability will be measured before and after the treatment through Quebec scale and Force Disability Scale Questionnaire in both groups.

DETAILED DESCRIPTION:
Groin pain mostly occurs in the first and second trimesters of pregnancy due to round ligament pain because the womb expands and causes stretching of ligaments making it more likely to become strained. The study will be focused on the effects of active tissue release techniques on groin pain, hip range of motion, and functional disability in 2nd trimester of pregnancy. A baseline treatment of ice therapy will be given for 10 minutes to all participants of this study. A sample of 30 will be divided into 2 groups. Group A will undergo treatment of active release techniques for 10 minutes thrice a week with no home plan of home relaxation exercises. In contrast, Group B will combine treatment of active release technology with home relaxation exercises.

Treatment will be given for 4 weeks and pain will be assessed before and after the treatment through (NPRS) scale. Functional disability will be measured before and after the treatment through the Quebec scale and Force Disability Scale Questionnaire in both groups. Recorded values will be analyzed for any change using SPSS

ELIGIBILITY:
Inclusion Criteria:

* Pain in the groin area/ Round Ligament pain
* NPRS scores between 4 to 10
* Functional activities scoring between 50 to 90 at Quebec score

Exclusion Criteria:

* Any diagnosed pathology like infection , malignancy ,inflammation
* Any structural deformity of lumbar and pelvic girdle,
* Any inguinal or lumbar surgery
* High risk pregnancy

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 4 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes. Changes from Baseline to 4 week.
The Quebec questionnaire: | up to 4 weeks
  The Quebec questionnaire is a condition-specific questionnaire developed to measure the level of functional disability for patients with groin pain. The original purpose of the questionnaire is to take into account the functional limitations related to pain, to monitor the progress of individual patients and to compare the evolution of groin pain subjects incorporated in rehabilitation programs
Goniometer: To measure range of motion: | up to 4 weeks
  A goniometer is a device that measures an angle or permits the rotation of an object to a definite position the range of motion is the measurement of movement around a specific joint or body part.

CONTACTS AND LOCATIONS:
Overall Officials: Khadija shamas, MS*, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Prime Care Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shiri R, Coggon D, Falah-Hassani K. Exercise for the prevention of low back and pelvic girdle pain in pregnancy: A meta-analysis of randomized controlled trials. Eur J Pain. 2018 Jan;22(1):19-27. doi: 10.1002/ejp.1096. Epub 2017 Sep 4. PMID 28869318
- [Background] Weir A, Jansen JA, van de Port IG, Van de Sande HB, Tol JL, Backx FJ. Manual or exercise therapy for long-standing adductor-related groin pain: a randomised controlled clinical trial. Man Ther. 2011 Apr;16(2):148-54. doi: 10.1016/j.math.2010.09.001. Epub 2010 Oct 16. PMID 20952244
- [Background] Cotellessa F, Puce L, Formica M, May MC, Trompetto C, Perrone M, Bertulessi A, Anfossi V, Modenesi R, Marinelli L, Bragazzi NL, Mori L. Effectiveness of a Preventative Program for Groin Pain Syndrome in Elite Youth Soccer Players: A Prospective, Randomized, Controlled, Single-Blind Study. Healthcare (Basel). 2023 Aug 22;11(17):2367. doi: 10.3390/healthcare11172367. PMID 37685401
- [Background] Andrews CM, O'Neill LM. Use of pelvic tilt exercise for ligament pain relief. J Nurse Midwifery. 1994 Nov-Dec;39(6):370-4. doi: 10.1016/0091-2182(94)90156-2. PMID 7830145
- [Background] Liddle SD, Pennick V. Interventions for preventing and treating low-back and pelvic pain during pregnancy. Cochrane Database Syst Rev. 2015 Sep 30;2015(9):CD001139. doi: 10.1002/14651858.CD001139.pub4. PMID 26422811
- [Background] Hall H, Cramer H, Sundberg T, Ward L, Adams J, Moore C, Sibbritt D, Lauche R. The effectiveness of complementary manual therapies for pregnancy-related back and pelvic pain: A systematic review with meta-analysis. Medicine (Baltimore). 2016 Sep;95(38):e4723. doi: 10.1097/MD.0000000000004723. PMID 27661020